CLINICAL TRIAL: NCT06254716
Title: A Retrospective Single-center Cohort Study on the Prognosis of Disc Resection and Segmental Resection Followed by Anastomosis on Gastrointestinal Function and Quality of Life in Patients With Rectal Endometriosis
Brief Title: A Study on the Prognosis of Two Different Surgery Methods in Patients With Rectal Endometriosis
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhang Wei, professor, Fudan University
Other Study IDs: FudanU2024-01-17
Record Dates: First submitted 2024-01-17; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Gastrointestinal Function; Quality of Life; Pregnancy Outcomes
Keywords: rectal endometriosis; disc resection; segmental resection; anastomose; gastrointestinal function
MeSH Terms: interventions — Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Disc resection of rectal endometriosis: Patients who underwent disc resection and anastomosis for rectal endometriosis involving the full thickness of the rectum reaching the mucosa or submucosa during preoperative evaluation or intraoperative exploration, and who were diagnosed pathologically.
  Interventions: Procedure: disc resection
- Segmental resection of rectal endometriosis: Patients who underwent segmental resection and anastomosis for rectal endometriosis involving the full thickness of the rectum reaching the mucosa or submucosa during preoperative evaluation or intraoperative exploration, and who were diagnosed pathologically.
  Interventions: Procedure: segmental resection

INTERVENTIONS:
Procedure: disc resection — disc resection refers to the full-thickness resection of the lesion and the intestinal wall, usually anterior rectal wall. During the operation, the anterior intestinal wall is opened and then sutured or anastomosed with a stapler. Segmental bowel resection for the treatment of intestinal endometriosis was first reported by Redwine and Sharpe in 1991, which requires the maximum removal of endometriosis lesions.
  Groups: Disc resection of rectal endometriosis
Procedure: segmental resection — Segmental bowel resection for the treatment of intestinal endometriosis was first reported by Redwine and Sharpe in 1991, which requires the maximum removal of endometriosis lesions.
  Groups: Segmental resection of rectal endometriosis

SUMMARY:
This retrospective study aims to compare the surgical and pregnancy outcomes of disc and segmental resection for rectal DIE through a single-center retrospective analysis, to summarize clinical experience, and to explore the possible factor of the differences. The results would provide preliminary clinical basis for the treatment and selection of surgical methods for patients with rectal DIE, and also provide a research basis for the prospective clinical studies.

DETAILED DESCRIPTION:
1. Research objectives This study aims to compare the surgical and pregnancy outcomes of disc and segmental resection for rectal DIE through a single-center retrospective analysis, to summarize clinical experience, to explore the possible factor of the differences and to followed up on the fertility outcomes of those who desire for pregnancy. The results would provide preliminary clinical basis for the treatment and selection of surgical methods for patients with rectal DIE, and also provide a research basis for the prospective clinical studies.
2. Innovation points In this retrospective study, innovation points are to compare the disease relief, perioperative complications and recurrence of two different surgical methods, disc resection and segmental resection, for rectal DIE involving the rectal mucosa and submucosa, and summarize past clinical experience. In order to provide preliminary clinical basis for the treatment and selection of surgical methods for patients with rectal DIE.
3. Research the main content This project intends to conduct a retrospectively observational study to collect the clinical data of patients with rectal DIE who underwent disc resection and segmental resection in a single center, to analyze perioperative complications, and to follow up the patients' symptom relief and recurrence. For those who desire for fertility, follow up their fertility status and pregnancy outcomes. By summarizing past clinical experience and exploring the possible influencing factors of the differences, we hope to provide preliminary clinical basis for the treatment and selection of surgical methods for patients with rectal DIE.
4. Key research methods and technologies:

Research methods: Single-center retrospective study

1. Case collection: Collect patients who were hospitalized in the Obstetrics and Gynecology Hospital of Fudan University in Shanghai from 2018 to 2023 and received surgical treatment for rectal endometriosis.

   Inclusion criteria: Patients who underwent surgery for endometriosis and were found to have endometriosis involving the full thickness of the rectum reaching the mucosa or submucosa during preoperative evaluation or intraoperative exploration, and who were diagnosed pathologically.

   Exclusion criteria: patients who have previously undergone surgical treatment of rectal endometriosis; patients with insufficient preoperative evaluation (lack of pelvic imaging evaluation or colonoscopy evaluation) and surgical removal of lesions; postoperative pathology shows rectal mucosa or The submucosa is not involved; patients with malignant tumors.
2. Case information collection: patient age, body mass index, menstrual status (menstrual period, cycle, menstrual volume), reproductive history, pain symptoms and extent (dysmenorrhea, dyspareunia), intestinal symptoms (constipation, diarrhea, anal incontinence and blood in the stool) , history of infertility, polycystic ovary syndrome, abdominal surgery history (number of surgeries and endometriosis-related surgeries), imaging evaluation (ultrasound and magnetic resonance evaluation results: adenomyosis, ovarian uterus Endometriosis cysts, organs involved in deep endometriosis, location, size, number, depth of rectal lesions and circumference of the intestinal tube involved), colonoscopy evaluation results, preoperative hormone treatment status and time (GnRHa , oral short-acting contraceptives, Mirena, dienogest, progesterone, etc.), tumor markers (CA125, CA199, CEA, etc.), AMH and preoperative hemoglobin, surgical methods (open, traditional laparoscopy, single hole laparoscopy), surgical method of rectal lesion resection (butterfly resection and segmental resection), anastomosis method (suture, stapler), distance from the lesion to the anus, size of the resected lesion (diameter, depth and circumference) , surgical content (hysterectomy, ovarian resection, and other endometriosis surgeries), operation time and amount of bleeding.
3. Surgical outcomes: decrease in hemoglobin, postoperative fever (whether ≥38°C), postoperative infection (pathogens confirmed by culture), perioperative blood transfusion treatment, postoperative complications (rectovaginal fistula, anastomotic fistula, Pelvic hematoma, urinary retention, organ damage, bleeding and multiple surgeries), postoperative hospitalization time, pathology (diameter, depth and circumference), postoperative auxiliary medication regimen and time (GnRHa, oral short-acting contraceptive pills , Mirena, dienogest, progesterone, etc.).
4. Pregnancy-related: whether there is a desire to get pregnant; the time to prepare for pregnancy after surgery; whether there are male infertility factors; pregnancy outcomes (pregnancy interval, natural conception rate, assisted reproduction pregnancy rate, miscarriage rate, pregnancy rate).
5. Recurrence: symptom assessment (pain level using VAS score and intestinal function recovery: frequency of defecation, stool shape, defecation pain, defecation effort) and imaging recurrence (magnetic resonance imaging shows lesions in the rectum).
6. Follow-up method: Obtain preliminary results through outpatient electronic medical records; telephone follow-up for patient symptom assessment.
7. Data analysis: Use SPSS software for data analysis. In descriptive statistics, categorical variables are expressed as numbers (percentages), and continuous variables are expressed as mean ± standard deviation. The t test was used to compare continuous variables between groups with normal distribution; the Mann-Whitney U test was used to compare continuous variables between groups with skewed distribution; the chi-square test was used to compare categorical variables between groups. The K-M curve plots postoperative recurrence and postoperative pregnancy. p<0.05 is considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent surgery of disc and segmental resection followed by anastomosis for endometriosis
* Endometriosis involving the full thickness of the rectum reaching the mucosa or submucosa during preoperative evaluation or intraoperative exploration, and who were diagnosed pathologically.

Exclusion Criteria:

* Patients who have previously undergone surgical treatment of rectal endometriosis
* Patients with insufficient preoperative evaluation (lack of pelvic imaging evaluation or colonoscopy evaluation) and surgical removal of lesions;
* Postoperative pathology shows rectal mucosa or The submucosa is not involved; patients with malignant tumors.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Patient age, body mass index, menstrual status (menstrual period, cycle, menstrual volume), reproductive history, pain symptoms and extent (dysmenorrhea, dyspareunia), intestinal symptoms (constipation, diarrhea, anal incontinence and blood in the stool) , history of infertility, polycystic ovary syndrome, abdominal surgery history (number of surgeries and endometriosis-related surgeries), imaging evaluation (ultrasound and magnetic resonance evaluation results: adenomyosis, ovarian uterus Endometriosis cysts, organs involved in deep endometriosis, location, size, number, depth of rectal lesions and circumference of the intestinal tube involved), colonoscopy evaluation results
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
complication rate of surgery | one year after surgery
  rate of rectovaginal fistula or anastomotic fistula
gastrointestinal function | one year after surgery
  The scoring of lower anterior resection syndrome (lower anterior resection syndrome
recurrence rate | one year after surgery
  Recurrence rate of symptoms or image findings

SECONDARY OUTCOMES:
gastrointestinal function- related quality of life index | one year after surgery
  gastrointestinal function- related quality of life index, Gastrointestinal function- related quality of Life Index, GIQLI, visual analogue scale (VAS) and endometriosis health profile (EHP-30).
pregnancy outcome | one year after surgery
  natural conception rate

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, Ph.D., Study Director — OB & GYN Hospital of Fudan University
Locations (1):
- OB & GYN Hospital of Fudan University, Shanghai, Shanghai Municipality, China